CLINICAL TRIAL: NCT01398878
Title: Assessing the Impact of a Change to the Work Schedule of Resident Physicians: a Mixed Methods Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Michael Smith Foundation (Unknown)
Responsible Party: Dr. Najib Ayas, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: H09-02007
Record Dates: First submitted 2011-07-11; First posted 2011-07-21 (Estimated); Last update posted 2011-07-25 (Estimated); Status verified 2011-07

CONDITIONS: Patient Safety; Resident Work Hours
Keywords: Medical education, graduate; Patient care; Outcome assessment (Health care); Work schedule tolerance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Traditional work schedule (No Intervention): Residents in the intensive care unit perform overnight shifts in excess of 24 hrs every fourth night
- Intervention work schedule (Active Comparator): Residents in the Intensive Care Unit perform shifts less than 16 hours in length and have at least 8 hours off between shifts
  Interventions: Behavioral: Intervention work shift

INTERVENTIONS:
Behavioral: Intervention work shift — Shiftwork schedule with elimination of shifts greater than 16 hours in length and at least 8 hours off between shifts for all residents in the Intensive Care Unit
  Arms: Intervention work schedule

SUMMARY:
The purpose of this study is to determine the impact of eliminating traditional resident work shifts (i.e. greater than 24 hours in length) on patient safety and resident educational outcomes. In addition, the investigators will explore with key stakeholders (patients and their families, nurses, resident physicians and attending physicians) their experiences when residents are undertaking shifts greater than 24 hours in length as compared to 16 hours or less.

ELIGIBILITY:
Inclusion Criteria:

* Residents completing Intensive Care Unit rotations
* For focus groups and interviews, patients and families members admitted during the study period and nurses and attending physicians working during the study period

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2011-07; Primary Completion 2012-06 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Preventable adverse events | Occurring during course of ICU admission and within first 72 hours of ICU discharge if event is attributable to process of care in the ICU
  The primary outcome is the rate of preventable adverse events per 1000 patient days. An adverse event will be defined as any unplanned injury arising as a consequence of medical care that is associated with morbidity, requires treatment, prolongs hospital stay, or results in disability at discharge. Adverse events are not caused by the disease process itself, but do include any procedural or therapeutic complications. Preventable adverse events will be defined as those adverse events that could have been avoided given current knowledge and standards of care.

SECONDARY OUTCOMES:
Quantity of scheduled and unscheduled learning activities residents participate in | End of each 28 day rotation
  Assessed by review of sleep/activity log
Resident leisure time, sleep, and time spent in the hospital | End of each 28 day rotation
  Assessed by review of sleep/activity log
Professionalism | End of each 28 day rotation
  In order to further explore this qualitative outcome measure, during structured interviews of residents, attending physicians, nurses and patients and their families, specific questions will be used to probe the perceived level of resident professionalism. For example, degree of commitment and professional investment in individual patients, and degree of commitment to the profession of medicine.
Nursing impact | Over course of study (12 months)
  In order to further explore this qualitative outcome measure, during focus groups with nurses specific questions will be used to probe the perceived level of impact on nursing.
Attending physician workload | Over course of study (12 months)
  In order to further explore this qualitative outcome measure, during structured interviews of attending physicians specific questions will be used to probe the perceived level of physician workload. For example, the difference in level of direct involvement in patient care activities (writing notes, performing procedures, etc) between the two schedules.
Perceived continuity of care | Over course of study (12 months)
  In order to further explore this qualitative outcome measure, during structured interviews of residents, attending physicians, nurses and patients and their families, specific questions will be used to probe the perceived level of continuity of care.
Quality of life | End of each 28 day rotation
  In order to further explore this qualitative outcome measure, during structured interviews of residents specific questions will be used to probe the perceived level of quality of life for the different call schedules.
Resident knowledge acquisition and retention | End of each 28 day rotation
  Scores on validated multiple choice question exams
Patient satisfaction | Within two weeks of ICU discharge
  Given the multitude of potential variables that impact patient satisfaction, during the interviews of patients and their families, the following questions will be used to inform the outcome measure: a global assessment of the patient's experience, their satisfaction with the overall care provided by the healthcare team and their satisfaction with their experiences with resident physicians in particular.
Job satisfaction/Stress | End of each 28 day rotation
  In order to further explore this qualitative outcome measure, during structured interviews of residents specific questions will be used to probe the perceived level of job satisfaction and stress for the different call schedules.

CONTACTS AND LOCATIONS:
Overall Officials: Najib Ayas, MD MPH, Principal Investigator — University of British Columbia
Locations (1):
- St Paul's Hospital, Vancouver, British Columbia, Canada